CLINICAL TRIAL: NCT05841550
Title: A Phase 1/Phase 2 Study to Investigate Safety, Tolerability and Efficacy With TG01/QS-21 Vaccine Administration in Patients With Confirmed KRAS or NRAS Codon 12/13 Mutation and High-risk Smoldering Multiple Myeloma or Multiple Myeloma and Evidence of Measurable Disease ≥ 1 Line of Treatment
Brief Title: The TG01 Study With TG01/QS-21 Vaccine in Patients With High-risk Smouldering Multiple Myeloma and Multiple Myeloma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Targovax ASA (Industry)
Responsible Party: Principal Investigator, Fredrik Hellem Schjesvold, Principal Investigator, Head of Oslo Myeloma Center, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OMC04
Record Dates: First submitted 2023-03-13; First posted 2023-05-03 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Multiple Myeloma; Smoldering Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma; Smoldering Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TG01 (Experimental): TG01 is a sterile lyophilizate consisting of a mixture of seven peptides. The finished product is a white powder for injection, consisting only of the active substances containing 2.1 mg of peptides (individual peptides comprising 0.3 mg each). The lyophilizate is to be reconstituted with QS-21 for injection before use.
  QS-21 is a naturally occurring saponin molecule purified from the South American tree Quillaja saponaria Molina. QS-21 Solution is supplied in a 2 mL CZ resin vial as a sterile, solution in PBS (phosphate buffered saline) at a concentration of 0.5 mg/mL QS-21 (500 mcg/mL) with each vial containing 0.7 mL intended single use only.
  The vaccine will be given subcutaneously Treatment consists of 12 doses TG01/QS-21 vaccine given every 2 weeks in the first 12 weeks, followed by every 8 weeks until week 52.
  TG01 dose 0.7 mg dose and QS-21 50 ug.
  Interventions: Biological: TG01

INTERVENTIONS:
Biological: TG01 — All participants will receive the same treatment as described under arm

SUMMARY:
The goal of this clinical trial is to test the safety, tolerability, and efficacy of TG01 vaccination in patients with KRAS or NRAS mutation on codon 12/13 mutation who has multiple myeloma or high-risk smoldering multiple myeloma. The main question it aims to answer are:

Is TG01/QS-21 vaccination safe and tolerable for this patient group? Is TG01/QS-21 vaccination treatment efficient in this group in terms of increased overall response rate, overall survival rate, progression-free survival, and time til next treatment? Is there an immunological response to the vaccine? Participants will be given TG01/QS-21 vaccination treatment. Treatment consists of 12 doses of TG01/QS-21 vaccine given every two weeks in the first 12 weeks, followed by every eight weeks until week 52.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 18 years of age
* RAS mutation (KRAS/NRAS codon 12/13 mutation) detected on archival or fresh bone marrow material with VariantPlex Myeloid Panel
* Confirmed diagnosis of high-risk smoldering multiple myeloma (SMM) according to IMWG criteria (30) and high-risk criteria as listed up below OR confirmed diagnosis of multiple myeloma (MM) according to IMWG criteria and measurable disease following ≥

  1 line of treatment
* In patients with high-risk SMM at least 2 of 3 following abnormalities, based on laboratory data obtained at screening must be fulfilled:

  1. Serum M-protein >20 g/L.
  2. Serum involved/uninvolved FLC ratio >20.
  3. BMPC >20%. OR presence of ≥10% BMPC and at least one of the following based on laboratory data obtained at screening:

     * Serum M-protein ≥30 g/L (If IgA, IgA ≥20g/L)
     * Serum involved/uninvolved FLC ratio ≥8 (but <100)
     * Abnormal PC immunophenotype (≥95% of BMPCs are clonal) and reduction of ≥1uninvolved Ig isotype (Only IgG, IgA and IgM will be considered)
     * Progressive increase in Serum M-protein level (evolving type of SMM) defined as an increase of Serum M-protein ≥10% in the last 12 months before enrolment in the study. This increase must be consistent from one to another sample (i.e., no decrease observed between 2 increased Serum M-protein values)
* Both high-risk SMM and MM patients must have evidence of measurable disease in accordance with IMWG criteria
* If patient with MM was eligible for ASCT, ASCT must have been performed, and patients cannot be enrolled until 3 months after ASCT
* Patient should not be expected to require immediate, subsequent line of treatment for at least 2 months
* Patient has not had reduction of clonal plasma cell markers for last two cycles (last two months if off treatment). If a patient had no reduction during the last two cycles of induction before ASCT, the patient can be enrolled, provided 3 months after ASCT
* Following ASCT, the patient cannot be enrolled without having tried lenalidomide maintenance given at standard doses for at least two cycles, if the clonal markers had a reduction during the last 2 cycles of induction treatment. Lenalidomide will be stopped when entering the study
* ECOG performance status 0-1
* Female patients of child-bearing potential (FCBP) must have negative serum pregnancy test at Screening and agree to use a highly effective method of contraception during treatment and for 3 months following last dose of drug.
* Male patients must use an effective barrier method of contraception during treatment and for 3 months following the last dose if sexually active with a FCBP.
* Ability to provide written informed consent and can understand and comply with the requirements of the study

Exclusion Criteria:

* Pregnant or lactating women or women without a pregnancy test at baseline (postmenopausal women must have been amenorrhoeic for at least 12 months to be considered of non-childbearing potential)
* Medical conditions such as but not limited to:

  1. Any uncontrolled infection
  2. Uncontrolled cardiac failure classification III or IV (NYHA)
  3. Uncontrolled systemic and gastro-intestinal inflammatory conditions
  4. History of adverse reactions to vaccines
* Active malignancy with worse prognosis than multiple myeloma
* Likely to require treatment intervention for multiple myeloma within two months of start of treatment with TG01/QS-21
* Known history of positive tests for HIV/AIDS, hepatitis B or C
* Planned to receive yellow fever or other live (attenuated) vaccines during the course of study
* Known hypersensitivity to QS-21.
* Only participants who are able to consent will be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-05-19 (Actual); Primary Completion 2027-05-19 (Estimated); Study Completion 2035-05-19 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with adverse events (AEs) | Baseline until 30 days after last dose of study drug, up to approximately 3 years
  An Adverse Event is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Percentage of participants discontinuing treatment secondary to treatment-related adverse events | Up to approximately 3 years
  Percentage of participants discontinuing treatment secondary to treatment-related adverse events

SECONDARY OUTCOMES:
Number of patients with Progression Free Survival (PFS) | Baseline to 11 years
  defined as the time from study treatment start to disease progression for every patient
Concentration of TG01-specific T-cell specific cytokine production | Baseline until end of study, assessed up to 11 years
  The immune response to TG01 will be measured by IFNg/TNFa ELISPOT or FluoroSpot quantifying the TG01 T-cell specific cytokine production. A positive immune response will be defined as a 2-fold higher mean spot number in experimental wells (with vaccine peptides) compared to control wells (medium)
Overall response rate per patient | Baseline to approximately 3 years
  The proportion of patients who achieve partial response (PR) or better following at least one dose of study treatment
Overall Survival (OS) per patient | Baseline until the end of study, assessed up to 11 years
  The OS rate of patients receiving 1 or more study treatments
Time to next treatment (TTNT) per patient | Baseline until the end of study, assessed up to 11 years
  defined as the time between the start date of the current treatment line and the start date of the next treatment line

CONTACTS AND LOCATIONS:
Overall Officials: Fredik Schjesvold, MD PhD, Principal Investigator — Oslo Myeloma Center, Oslo University Hospital
Locations (1):
- Oslo Myeloma Center, Oslo, Oslo County, Norway

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, Informed consent form, Clinical trial results, Investigator Brochure, IMPD
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Study protocol, Informed consent form immediate after trial is approved. Clinical trial results summary and lay person summary 12 months after end of trial date. Clinical trial results summary for an intermediate data analysis 12 months after interim data analysis date. IMPD SandE sections and Investigator Brochure 7 years after end of trial.
Access Criteria: Anyone who wish access to the data